CLINICAL TRIAL: NCT06283212
Title: EXPEDITION: A Clinical Study to Evaluate the Safety and Efficacy of ETX101, an AAV9-Delivered Gene Therapy in Children With SCN1A-positive Dravet Syndrome
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of ETX101, an AAV9-Delivered Gene Therapy in Children With SCN1A-positive Dravet Syndrome
Acronym: UK Only
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Encoded Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETX-DS-005
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Cohort A will evaluate ETX101 dose level 1.
  Interventions: Drug: ETX101
- Cohort B (Experimental): Cohort B will evaluate ETX101 dose level 2.
  Interventions: Drug: ETX101
- Cohort C (Experimental): Cohort C will evaluate ETX101 dose level 3.
  Interventions: Drug: ETX101
- Cohort D (Experimental): Cohort D will evaluate ETX101 dose level 4.
  Interventions: Drug: ETX101

INTERVENTIONS:
Drug: ETX101 — ETX101 is composed of a non-replicating, recombinant adeno-associated viral serotype 9 (rAAV9) vector used to deliver a GABAergic regulatory element (reGABA) and an engineered transcription factor that increases transcription of the SCN1A gene (eTFSCN1A)

SUMMARY:
EXPEDITION is a Phase 1/2 study in the UK to evaluate the safety and efficacy of ETX101 in participants with SCN1A-positive Dravet Syndrome aged 6 to < 48 months. The study follows and open-label, dose-escalation design.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a predicted loss of function pathogenic or likely pathogenic SCN1A variant
* Participant must have experienced their first seizure between the age of 3 and 15 months
* Participant must have a clinical diagnosis of Dravet syndrome or the treating clinician must have high clinical suspicion of a diagnosis of Dravet syndrome
* Participant is receiving at least one prophylactic antiseizure medication

Exclusion Criteria:

* Participant has another genetic mutation or clinical comorbidity which could potentially confound the typical Dravet phenotype
* Participant has a known central nervous system structural and/or vascular abnormality (indicated by an MRI or CT scan of the brain).
* Participant has an abnormality that may interfere with CSF distribution and/or has an existing ventriculoperitoneal shunt.
* Participant is currently taking or has taken antiseizure medications (ASMs) at a therapeutic dose that are contraindicated in Dravet syndrome, including sodium channel blockers.
* Participant has experienced seizure freedom for a period of 4 consecutive weeks within the 90-day period prior to informed consent.
* Participant has previously received gene or cell therapy.
* Participant is currently enrolled in a clinical trial or receiving an investigational therapy.
* Participant has clinically significant underlying liver disease.

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Proportions of participants experiencing any treatment-emergent adverse events (AEs), serious adverse events (SAEs), related AEs, AEs with severity Grade ≥ 3, AEs resulting in study discontinuation, and AEs with fatal outcome. | Day 1 through Study Completion, an average of 5 years
Change from baseline in the standard score of the Vineland Adaptive Behavior Scales - Third Edition Adaptive Behavior Composite at Week 52. | Baseline to Week 52. Standard scores are normalized to a mean and SD of 100 and 15, respectively, and are not bounded by a range. Higher scores correspond to better outcomes.

SECONDARY OUTCOMES:
Percent change in monthly countable seizure frequency (MCSF) to Week 52, with countable seizures defined as generalized tonic-clonic/clonic, focal motor with clearly observable clinical signs, tonic bilateral, and atonic seizures. | Between the 8-week baseline period and the 48-week post-dosing assessment period (defined as Week 5 to Week 52 following administration of ETX101)
Change from baseline in the raw score of the Bayley Scales of Infant and Toddler Development® 4th Edition receptive language sub-domain at Week 52. | Baseline to Week 52. Raw scores range from 0 to 49 and higher scores correspond to better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Rico, M.D., Ph. D, Study Director — Encoded Therapeutics
Locations (3):
- United Kingdom (3):
  - Queen Elizabeth Hospital, Glasgow
  - Great Ormond Street Hospital, London
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No